CLINICAL TRIAL: NCT00923663
Title: Phase II Trial of Lenalidomide in Patients With Lymphoma of the Mucosa Associated Lymphoid Tissue (MALT) Type
Brief Title: Trial of Lenalidomide in Patients With Lymphoma of the Mucosa Associated Lymphoid Tissue (MALT) Type
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof Markus Raderer, Internal Medicine I, Division of Oncology, University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEN-MALT
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: MALT Lymphoma
Keywords: MALT lymphoma; Advanced or Helicobacter pylori-refractory MALT lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Lenalidomide

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide administered orally at a dose of 25 mg daily
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 25 mg Lenalidomide p.o. daily for 21 days

SUMMARY:
The activity of monotherapy with Lenalidomide will be evaluated in patients with lymphoma of the mucosa associated lymphoid tissue (MALT).

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the clinical potential of Lenalidomide to induce objective/histologic responses in patients with MALT lymphoma.

The secondary objectives are to evaluate the safety of Lenalidomide in this patient population and to evaluate the impact of Lenalidomide on progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed MALT lymphoma with measurable disease (stage I - IV)
* With first or greater relapse after HP-eradication, radiation or chemotherapy in case of gastric lymphoma
* Age > 18 years
* Must be able to tolerate therapy, and have adequate cardiac, renal, and hepatic function, ECOG status of 0 - 2
* Must be capable of understanding the purpose of the study and have given written informed consent

Exclusion Criteria:

* Lymphoma histology other than MALT lymphoma or MALT lymphoma with a diffuse large cell lymphoma ("high grade lymphoma") - component
* Use of any investigational agent within 28 days prior to initiation of treatment with lenalidomide
* History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of the cervix within the last 5 years
* Major surgery, other than diagnostic surgery, within the last 4 weeks
* Evidence of CNS involvement
* A history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs
* Severe peripheral polyneuropathy
* Clinically significant cardiac disease (e.g., congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 6 months
* Inadequate hematological status at baseline prior to study entry: Dependency on red blood cell and/or platelet transfusions, ANC (absolute neutrophil count (segmented + bands)) < 1.0 x 109/L
* Patients with active opportunistic infections
* Pregnancy
* Uncontrolled diabetes mellitus
* Preexisting thromboembolic events at start of study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Rate of objective responses induced by Lenalidomide | 24 months

SECONDARY OUTCOMES:
Time to progression | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Internal Medicine, Vienna, Austria

REFERENCES:
- [Derived] Kiesewetter B, Troch M, Dolak W, Mullauer L, Lukas J, Zielinski CC, Raderer M. A phase II study of lenalidomide in patients with extranodal marginal zone B-cell lymphoma of the mucosa associated lymphoid tissue (MALT lymphoma). Haematologica. 2013 Mar;98(3):353-6. doi: 10.3324/haematol.2012.065995. Epub 2012 Aug 16. PMID 22899582